CLINICAL TRIAL: NCT04715646
Title: Open-Label, Single-Arm, Multicenter Study to Evaluate Long-Term Safety and Tolerability of Brivaracetam Used as Adjunctive Treatment in Pediatric Study Participants With Epilepsy
Brief Title: A Study to Test the Safety and Tolerability of Brivaracetam in Children and Adolescents With Seizures
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0156; 2020-003664-29 (EudraCT Number)
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Pediatric; Child
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brivaracetam (Experimental): LTFU study participants: Up to 5mg/kg/day (for study participants weighing 11kg to less than 20kg) and up to 4mg/kg/day (for study participants weighing 20kg to less than 50kg) and no more than 200mg/day Directly enrolled (DE) study participants: 1mg/kg/day to 4mg/kg/day and no more than 200mg/day.
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — Brivaracetam (BRV) tablets or oral solution will be administered twice daily (bid) in 2 equally divided doses.
  Tablet strengths: 10 mg, 25 mg, 50 mg Route of administration: oral
  Oral solution Concentration: 10 mg/ml Route of administration: oral
  Other Names: BRV; Briviact

SUMMARY:
The purpose of the study is to evaluate the long-term safety and tolerability of brivaracetam.

DETAILED DESCRIPTION:
EP0156 is designed to assess the long-term safety and tolerability of BRV in pediatric study participants with epilepsy who participated in the neonatal study N01349 [NCG03325439] and/or have participated in the open-label, long-term, follow-up pediatric study N01266 [NCT01364597]. EP0156 will also assess the long-term safety and tolerability of BRV in Japanese pediatric study participants with partial-onset seizures who will be directly enrolled into the study in Japan. Pharmacokinetic data will also be evaluated in Japanese study participants.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for long-term follow-up (LTFU) study participants only

* Study participants ≥ 1 month of age with a confirmed diagnosis of epilepsy who participated in core study N01266 [NCT01364597] and/or N01349 [NCT03325439]

Inclusion criteria for directly enrolled (DE) study participants in Japan only

* Study participant is ≥ 4 years to < 16 years of age
* Study participant has presence of an electroencephalogram (EEG) reading compatible with the diagnosis of focal epilepsy within the last 10 years
* Study participant has uncontrolled partial-onset seizure (POS) after an adequate course of treatment with at least 1 antiepileptic drug (AED)
* Study participant had at least 1 POS during the 4-week Screening Period

Exclusion Criteria:

Exclusion criteria for all study participants

* Severe medical, neurological, or psychiatric disorders or laboratory values, which may have an impact on the safety of the study participant
* Study participant is currently participating in another study of an investigational medication (or a medical device) other than brivaracetam (BRV).

Exclusion criteria for long-term follow-up (LTFU) study participants only

- Study participant ≥ 6 years of age has a lifetime history of suicide attempt or has suicidal ideation in the past 6 months as indicated on the Columbia Suicide Severity Rating Scale (C-SSRS)

Exclusion criteria for directly enrolled (DE) study participants in Japan only

* Study participant has a history of primary generalized epilepsy, psychogenic non-epileptic seizures, or febrile seizures
* Study participant has a history of status epilepticus in the 30 days prior to the Screening Visit (ScrV) or during the Screening Period
* Study participant has any clinically significant illness
* Study participant has clinically significant laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results
* Study participant has a clinically significant ECG abnormality
* Study participant had major surgery within 6 months prior to the ScrV

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2030-07-08 (Estimated); Study Completion 2030-07-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) during the study | From Evaluation Visit (Day 1) until Safety Visits (up to 5 years)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug.
Incidence of treatment-emergent serious adverse events (SAEs) during the study | From Evaluation Visit (Day 1) until Safety Visits (up to 5 years)
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly or birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Incidence of treatment-emergent adverse events (TEAEs) leading to discontinuation of study drug during the study | From Evaluation Visit (Day 1) until Safety Visits (up to 5 years)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (36):
- United States (2):
  - Ep0156 259, Hawthorne, New York
  - Ep0156 237, Durham, North Carolina
- Ep0156 204, Leuven, Belgium
- Ep0156 240, Prague, Czechia
- Ep0156 207, Loos, France
- Ep0156 209, Freiburg im Breisgau, Germany
- Hungary (3):
  - Ep0156 210, Budapest
  - Ep0156 247, Budapest
  - Ep0156 232, Miskolc
- Ep0156 230, Roma, Italy
- Japan (19):
  - Ep0156 803, Bunkyō City
  - Ep0156 808, Chūō
  - Ep0156 800, Gifu
  - Ep0156 807, Hiroshima
  - Ep0156 815, Kodaira-shi
  - Ep0156 813, Kōshi
  - Ep0156 806, Kyoto
  - Ep0156 811, Nagoya
  - Ep0156 812, Niigata
  - Ep0156 817, Osaka
  - Ep0156 818, Ōbu
  - Ep0156 819, Ōmura
  - Ep0156 805, Sapporo
  - Ep0156 816, Sendai
  - Ep0156 809, Shimotsuke
  - Ep0156 814, Shizuoka
  - Ep0156 804, Tokyo
  - Ep0156 810, Yokohama
  - Ep0156 802, Yonago
- Mexico (3):
  - Ep0156 223, Aguascalientes
  - Ep0156 609, Culiacán
  - Ep0156 603, Guadalajara
- Poland (3):
  - Ep0156 406, Kielce
  - Ep0156 402, Krakow
  - Ep0156 401, Poznan
- Ep0156 248, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org